CLINICAL TRIAL: NCT02113891
Title: Treatment of Subclinical Antibody-mediated Acute Rejection in Kidney Transplant Recipients With the Complement Inhibitor Eculizumab.
Brief Title: Eculizumab Therapy for Subclinical Antibody-mediated Rejection in Kidney Transplantation
Acronym: TAMARCIN
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: disengagement of the sponsor Alexion Pharmaceuticals
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Alexion Pharmaceuticals, Inc. (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P101004
Record Dates: First submitted 2013-11-21; First posted 2014-04-15 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Subclinical Acute Antibody-mediated Rejection in Kidney Transplantation
Keywords: Antibody-mediated rejection; Complement blockade; Eculizumab; Kidney transplantation
MeSH Terms: interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Eculizumab (Experimental): Eculizumab will be given in addition to standard immunosuppression regimen (tacrolimus, mycophenalte mofeti, prednisone)
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Eculizumab induction: 900 mg IV every 7 days for 4 doses, a fifth 1200 mg dose 7 days later Eculizumab maintenance: 15 1200 mg doses every 14 days.
  (each patient will receive a total of 20 eculizumab doses during the whole treatment period from 3 month to 12 month post-transplant).
  Other Names: Soliris

SUMMARY:
Advances in renal transplantation have increased life-expectancy in patients with end-stage kidney disease. Conventional immunosuppressive drugs prevent efficiently early allograft losses due to T-cell mediated rejection. However, emerging data suggest that the majority of late kidney failures may be attributable to antibody-mediated rejection (AMR), which poorly responds to the currently available therapeutics. Complement-fixing donor-specific anti-HLA antibodies are associated with the worst outcome in keeping with the well-established role of the complement in AMR pathogenesis. Eculizumab, the first licenced complement blocker, has been found efficient in reducing the occurrence of AMR lesions in highly sensitized patients. A few reports also suggest that complement blockade may be of great value as salvage therapy for graft-threatening severe AMR. However, no information is available in the literature about the interest of complement blockade in curbing the progression of subclinical acute AMR to chronic AMR.

The purpose of this study is to determine whether complement blockade with eculizumab is effective and safe in the treatment of subclinical AMR in sensitized kidney transplant recipients.

Despite appropriate therapies, up to 75% of patients having received a renal transplant with preformed donor-specific antibody display subclinical AMR on their 3-month protocol biopsy. Subclinical AMR is defined by histological lesions of AMR concomitant with stable graft function. Moreover, the extent of these lesions at 3 month post-transplant correlates with the occurrence of irreversible scars and chonic antibody-mediated rejection on the 12-month biopsy.

This study aims to explore the efficacy and safety of eculizumab in patients exhibiting subclinical AMR on their 3 month-post-transplant biopsy, to reduce or even normalize microcirculation inflammation, and to prevent chronic rejection (transplant glomerulopathy) on the 12 month-screening biopsy. Eculizumab-treated patients will be compared with historical controls, matched for the lesions on the 3 month biopsy.

DETAILED DESCRIPTION:
Advance in renal transplantation for the treatment of patients with end-stage kidney failure have led to significant improvements in patient survival. T-cell directed immunotherapeutic agents are capable of preventing early allograft loss and represent the cornerstone of current maintenance immunosuppressive regimens. However, recent studies have pointed out that the majority (63%) of late kidney failures could be attributable to antibody-mediated rejection. Microcirculation inflammation (poly and mononuclear cells within glomerular and peritubular capillaries) correlates best with alloantibody-induced endothelial damages and complement-fixing anti-HLA antibodies, predicts evolution toward chronic antibody mediated rejection (transplant glomerulopathy), and is associated with a poor outcome. Microcirculation inflammation, the hallmark lesions of AMR, are frequently observed (75%) on screening biopsies performed in sensitized patients having received a renal transplant across a positive crossmatch due to preformed DSA, despite intensive prophylactic therapy (including polyclonal immunoglobulin, plasma exchanges and rituximab).

Altogether these findings underscore the need for innovative treatment to better control the humoral arm of chronic rejection in patients with donor-specific anti-HLA antibodies. Short-term eculizumab treatment might be a promising avenue. Complement blockade with eculizumab has been found efficient in reducing the occurrence of AMR lesions in highly sensitized patients. A few reports also suggest that complement blockade may be of great value as salvage therapy for graft-threatening severe AMR. However, no information is available in the literature about the efficacy of complement blockade in curbing the progression of subclinical AMR to chronic AMR.

The primary objectives of this study are:

• To determine the effectiveness of eculizumab in reducing durably alloantibody-induced microcirculation inflammation and preventing chronic microcirculation damages on 12-month screening biopsies.

The secondary objectives of this study are:

* To assess the effect of eculizumab on serum creatinine levels, amount of proteinuria, and measured and estimated Glomerular Filtration Rate (mGFR) between 3 and 12 months post-transplant.
* To determine the effectiveness of eculizumab in hampering the appearance of interstitial fibrosis and tubular atrophy (IF/TA), and dampening down alloantibody-induced accelerated arteriosclerosis on 1-year-post-transplant biopsy.
* Incidence of biopsy-proven antibody-mediated acute rejection (rise of creatinine value higher than 20% above the baseline value).
* To monitor DSA levels at 3, 6 and 12 months post-transplant with solid-phase assay (Luminex).
* To assess vital signs (such as systolic, diastolic blood pressure, heart rate, weight, temperature) and laboratory parameters at every eculizumab administration.
* To collect safety data on infections, cardiovascular events, and malignancies
* To monitor endothelial, platelet and leukocyte microparticles as well as endothelial cell progenitors
* To quantify the number of endothelial and NK expressed genes that correlate with AMR

This is an open-label exploratory study which evaluates eculizumab administration in sensitized patients with subclinical antibody-mediated rejection at 3 month-post-transplant. Ten patients fulfilling inclusion/exclusion criteria will be enrolled into the study and compared with 20 historical controls matched for the sensitization and histological lesions at 3 months. The patients enrolled in this study will be given eculizumab from 3 to 12 month post-transplant, according to the standard protocol in adults heavier than 40 kg (900 mg weekly for 4 weeks, 1200 mg for the fifth infusion and 1200 mg every other week thereafter).

Clinical and laboratory evaluations including vital signs and safety laboratory values will be monitored at predetermined time points.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 -75 years.
* Patients having received a kidney transplant from a living or deceased donor
* Patients with stable renal function
* Sensitized patient with at least one anti-HLA class II DSA (MFI > 1000) within the first 3 months.
* Adequate 3-month-protocol biopsy exhibiting microcirculation inflammation defined by glomerulitis Banff score (g) superior or egal 2 and /or peri-tubular capillaritis Banff score (ptc) superior or egal 2, AND the sum of scores g + ptc superior or egal 3.
* C4d positive staining on 3-month-protocol biopsy
* Adequate 3-month-protocol biopsy exhibiting limited scarred areas as defined as IF/TA score (ci + ct) inferior or egal 2 and no or minimal transplant glomerulopathy (cg inferior or egal 1)
* Patients who have given written informed consent to participate in all aspects of the study.
* Females of childbearing potential must have a negative pregnancy test within 48 hours prior to the first eculizumab administration.

Exclusion Criteria:

* Patients with known hypersensitivity to eculizumab or drugs with similar chemical structure.
* Patients having experienced and having been treated for an acute antibody-mediated rejection within the first 3 months post-transplant
* Patients with multi-organ transplant
* Female patients who are pregnant, lactating or of child bearing potential and not practicing an approved method of birth control.
* Patients with a known malignancy or history of malignancy other than excised basal or squamous cell carcinoma of the skin
* HBV, HCV or HIV-chronically infected patients
* Patients with evidence of severe liver disease, including abnormal liver profile (aspartate aminotransferase [AST], alanine aminotransferases [ALT] or total bilirubin > 3 times upper limit of normal at screening.
* Patients with current severe infection.
* Ongoing meningococcal infection
* Patient with systemic lupus erythematosus disease and / or anti-phospholipid antibodies
* Patients with any surgical or medical condition, which in the opinion of the investigator precludes enrollment in this trial
* Patients who live far from the transplant center and are unable to comply with all study visits.
* Long-term anticoagulation therapy or other contraindication to graft biopsies
* Positive BKV viremia during the first three months post-transplant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2017-07 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Microcirculation inflammation | 12-month screening biopsies
  Compare trajectories of g (0-3) and ptc (0-3) Banff scores
Transplant glomerulopathy | 12 month screening biopsies
  Compare trajectories of cg (0-3) Banff score
Microcirculation inflammation | 3 month screening biopsies
  Compare trajectories of g (0-3) and ptc (0-3) Banff scores
Transplant glomerulopathy | 3 month screening biopsies
  Compare trajectories of cg (0-3) Banff score

SECONDARY OUTCOMES:
Measured Glomerular Filtration Rate (Iohexol clearance) | 12 months post-transplant
  Compare trajectories of GFR change and percent GFR change between the study group and historiacl controls
Incidence of adverse effects | at 15 months post-transplant
  Monitoring of adverse events as well as evaluation of changes in laboratory parameters
Incidence of biopsy-proven acute rejection | at 12 months post-transplant
  graft biopsy for cause (rise in creatinine level…)
CH50 | at 15 months post-transplant (baseline, each infusion, study completion)
  Monitoring of eculizumab pharmacodynamic with an in vitro complement activity assay (CH50).
Endothelial Microparticles and Progenitors | Baseline, 1, 3, 6 and 9 months
  Number of endothelial and leukocyte-derived microparticules, as well as circulating endothelial progenitors as a biomarker of the graft endothelium insult.
Molecular diagnosis of AMR | 3 and 12-month post-transplant biopsy
  Compare trajectories of endothelial and NK expressed genes between the study group and historiacl controls
Donor Specific Antibody titers (Luminex SA) | 3 months post-transplant
  Monitor the persistence of DSA in the study group in comparison with historical controls.
Measured Glomerular Filtration Rate (Iohexol clearance) | 3 months post-transplant
  Compare trajectories of GFR change and percent GFR change between the study group and historiacl controls
Donor Specific Antibody titers (Luminex SA) | 12 months post-transplant
  Monitor the persistence of DSA in the study group in comparison with historical controls.
Donor Specific Antibody titers (Luminex SA) | 9 months post-transplant
  Monitor the persistence of DSA in the study group in comparison with historical controls.
Donor Specific Antibody titers (Luminex SA) | 6 months post-transplant
  Monitor the persistence of DSA in the study group in comparison with historical controls.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe LEGENDRE, MD, Study Director — Service de Transplantation Rénale, Hôpital Necker Université Paris Descartes 149 rue de Sèvres 75015 Paris, France

REFERENCES:
- [Background] Loupy A, Suberbielle-Boissel C, Hill GS, Lefaucheur C, Anglicheau D, Zuber J, Martinez F, Thervet E, Mejean A, Charron D, Duong van Huyen JP, Bruneval P, Legendre C, Nochy D. Outcome of subclinical antibody-mediated rejection in kidney transplant recipients with preformed donor-specific antibodies. Am J Transplant. 2009 Nov;9(11):2561-70. doi: 10.1111/j.1600-6143.2009.02813.x. Epub 2009 Sep 22. PMID 19775320
- [Background] Stegall MD, Diwan T, Raghavaiah S, Cornell LD, Burns J, Dean PG, Cosio FG, Gandhi MJ, Kremers W, Gloor JM. Terminal complement inhibition decreases antibody-mediated rejection in sensitized renal transplant recipients. Am J Transplant. 2011 Nov;11(11):2405-13. doi: 10.1111/j.1600-6143.2011.03757.x. Epub 2011 Sep 22. PMID 21942930
- [Background] Loupy A, Lefaucheur C, Vernerey D, Prugger C, Duong van Huyen JP, Mooney N, Suberbielle C, Fremeaux-Bacchi V, Mejean A, Desgrandchamps F, Anglicheau D, Nochy D, Charron D, Empana JP, Delahousse M, Legendre C, Glotz D, Hill GS, Zeevi A, Jouven X. Complement-binding anti-HLA antibodies and kidney-allograft survival. N Engl J Med. 2013 Sep 26;369(13):1215-26. doi: 10.1056/NEJMoa1302506. PMID 24066742
- [Background] Zuber J, Le Quintrec M, Krid S, Bertoye C, Gueutin V, Lahoche A, Heyne N, Ardissino G, Chatelet V, Noel LH, Hourmant M, Niaudet P, Fremeaux-Bacchi V, Rondeau E, Legendre C, Loirat C; French Study Group for Atypical HUS. Eculizumab for atypical hemolytic uremic syndrome recurrence in renal transplantation. Am J Transplant. 2012 Dec;12(12):3337-54. doi: 10.1111/j.1600-6143.2012.04252.x. Epub 2012 Sep 7. PMID 22958221